CLINICAL TRIAL: NCT04061369
Title: Establishing Short-term Protocols for Measuring Resting and Postprandial Energy Expenditure and Substrate Oxidation in a Whole Room Calorimeter
Brief Title: Energy Expenditure and Substrate Oxidation in a Whole Room Calorimeter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After Covid-19 pandemic, room calorimeter not functional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FL106
Record Dates: First submitted 2019-07-22; First posted 2019-08-19 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-08

CONDITIONS: Overweight; Obesity; Body Weight
Keywords: thermic effect of feeding; thermogenesis; calorimeter; fuel utilization
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: The study will be a randomized design that includes a volunteer receiving one of four test meals.
Who Masked: Outcomes Assessor
Masking Description: Both the investigator and the participant will be aware of the group assignment. The persons handling the data and statistics will not be aware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meal 1 (Experimental): Meal consisting of conventional foods that is low (20% of energy) in fat calories.
  Interventions: Other: Low fat meal
- Meal 2 (Experimental): Meal consisting of conventional foods that is moderate (40% of energy) in fat calories.
  Interventions: Other: Moderate fat meal
- Meal 3 (Experimental): Meal consisting of conventional foods that is high (60% of energy) in fat calories.
  Interventions: Other: High fat meal
- Meal 4 (Experimental): A liquid meal, similar to a "smoothie", that is high (60% of energy) in fat calories.
  Interventions: Other: High fat liquid meal

INTERVENTIONS:
Other: Low fat meal — Meal consisting of conventional foods that is low (20% of energy) in fat calories.
  Arms: Meal 1
Other: Moderate fat meal — Meal consisting of conventional foods that is moderate (40% of energy) in fat calories.
  Arms: Meal 2
Other: High fat meal — Meal consisting of conventional foods that is high (60% of energy) in fat calories.
  Arms: Meal 3
Other: High fat liquid meal — Liquid meal that is high (60% of energy) in fat calories.
  Arms: Meal 4

SUMMARY:
The investigators aim to establish a protocol for metabolic rate measurements obtained using continuous monitoring of oxygen consumption and carbon dioxide production in a whole room calorimeter setting.

DETAILED DESCRIPTION:
The purpose of this study is to determine the duration and time course of the thermic effect of single meals consumed by subjects who have been previously fasting for 12 hours overnight. Capturing the full thermic effect of a meal may take up to 8 hours, depending on the calorie load, nutrient composition of the meal, and rate of digestion. The investigators will test meals consisting of conventional foods that are low (20% of energy), moderate (40% of energy) or high (60% of energy) in fat calories, as fat is thought to slow the digestive process. The investigators will test a liquid meal, that is high (60% of energy) in fat calories, as liquid foods are thought to move more quickly through the digestive process. Another purpose of this study is to determine the test-retest reproducibility for the meals described above. To accomplish reproducibility, a volunteer will be permitted to repeat a test day two times using the same test meal.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 18.5 - 39.9 kg/m2

Exclusion Criteria:

* BMI < 18.5 or > 40 kg/m2
* Presence of untreated or uncontrolled metabolic diseases
* Presence of gastrointestinal distress or disorders that prevent consumption of a study meal (in particular, the high fat meals)
* Presence of Crohn's disease, irritable bowel syndrome, or colitis
* Previous gallbladder removal
* Presence of cancer or other serious chronic disease
* Implanted medical device that is battery operated, such as a pacemaker, defibrillator, electrocardiograph, or nerve simulator
* Presence of a large amount of metal in the body such as a hip implant
* Current use of tobacco in any form
* Claustrophobia
* Dietary restrictions that would interfere with consuming study meals
* Pregnant or nursing within the last 6 months, or plan to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Baseline level and change in rate of oxygen consumption | Measured continuously from baseline up to 600 minutes post-meal
  Oxygen consumption rate (VO2/min) measured by gas analyzer while inside whole room calorimeter
Baseline level and change in rate of carbon dioxide production | Measured continuously from baseline up to 600 minutes post-meal
  Carbon dioxide production rate (VCO2/min) measured by gas analyzer while inside whole room calorimeter
Baseline level and change in respiratory exchange ratio (RER) | Measured continuously from baseline up to 600 minutes post-meal
  RER is expressed as the ratio of VCO2 to VO2
Baseline level and change in urinary nitrogen excretion | Measured from discrete specimens and a pooled urine sample collected up to 600 minutes post-meal while in the room calorimeter
  Urinary nitrogen measured via combustion and gas analysis in mg

SECONDARY OUTCOMES:
Body weight | Baseline
  measured in kg
Body fat | Baseline
  Measured in kg using multi frequency bioimpedance
Lean body mass | Baseline
  Measured in kg using multi frequency bioimpedance
Total body water | Baseline
  Measured in kg using multi frequency bioimpedance
Waist circumference | Baseline
  measured in cm
Hip circumference | Baseline
  measured in cm
Blood pressure | Baseline
  Both systolic and diastolic pressure measured in mmHg using automated instrument
Heart rate | Baseline
  measured in beats per minute using automated instrument
Body temperature | Baseline
  measured in centigrade
General health and well-being | Baseline
  The SF-36 Short form general health and well-being questionnaire measured once. The survey has eight scales; physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health. All 36 items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Items in the same scale are averaged together to create the 8 scale scores.
Usual physical activity | Baseline
  Physical activity estimated from the Stanford Brief Physical Activity questionnaire. Scale is categorical for two subscales: work physical activity and leisure time activity.
Baseline level and change in satiety | Baseline, and 5, 10, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, and 480 minutes after meal
  Self-reported feelings of fullness measured on a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 100 or "extremely."
Baseline level and change in hunger | Baseline, and 5, 10, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, and 480 minutes after meal
  Self-reported feelings of hunger measured on a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 100 or "extremely."
Baseline level and change in desire to eat | Baseline, and 5, 10, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, and 480 minutes after meal
  Self-reported feelings of the desire to eat measured on a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 100 or "extremely."
Baseline level and change in prospective consumption | Baseline, and 5, 10, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, and 480 minutes after meal
  Self-reported feelings of prospective consumption measured on a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 100 or "extremely."
Baseline level and change in energy expenditure | Expressed from baseline up to 600 minutes post-meal
  Calculated as kcal/min from oxygen consumption and carbon dioxide production (L/min) and urinary nitrogen excretion (g/min)
Baseline level and change in carbohydrate combustion | Expressed from baseline up to 600 minutes post-meal
  Calculated as g/min from oxygen consumption and carbon dioxide production (L/min) and urinary nitrogen excretion (g/min)
Baseline level and change in fat combustion | Expressed from baseline up to 600 minutes post-meal
  Calculated as g/min from oxygen consumption and carbon dioxide production (L/min) and urinary nitrogen excretion (g/min)
Baseline level and change in thermic effect of food (TEF) | Expressed from baseline up to 600 minutes post-meal
  Calculated as the increase in post-meal energy expenditure above baseline energy expenditure
Baseline level and change in heart rate | Expressed from baseline up to 600 minutes post-meal
  Heart rate is estimated from wrist-worn activity monitor

CONTACTS AND LOCATIONS:
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No